CLINICAL TRIAL: NCT02181751
Title: A 1-year Program to Treat Children Who Have Been Victims of Child Sexual Abuse
Status: Withdrawn | Type: Observational
Why Stopped: Study was never initiated
Sponsor: Little Warriors (Other)
Responsible Party: Sponsor
Other Study IDs: LW2014
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Sexual Abuse of Child (If Focus of Attention is on Victim)
Keywords: Child Sexual Abuse; CSA; Treatment; Prevention; PTSD; Post Traumatic Stress Disorder; Depression; Anxiety; Quality of Life; Attachment; Cognitive Behavioural Therapy; Group Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment Group: Children in the Treatment Group will receive treatment for a Trauma Focused Cognitive Behavioural Therapy Group.
  Interventions: Other: Trauma Focused Cognitive Behavioural Therapy Group

INTERVENTIONS:
Other: Trauma Focused Cognitive Behavioural Therapy Group — Youth may participate in trauma focused cognitive behavioural group therapy (TF-CBT)

SUMMARY:
Our goal in this study is examine if a program designed to decrease the severity of Post-Traumatic Stress Disorder symptoms in sexually abused children between the ages of 8-12 was effective.

ELIGIBILITY:
Inclusion Criteria:

* History of sexual abuse
* Aged 8 - 12 years
* Developmentally able to be on-site in a "camp-like" treatment facility for 3 weeks with their parent/guardian (or without if family is not available to join the child at the Be Brave Ranch)
* Able to perform skills of daily living for self care
* Good physical health

Exclusion Criteria:

* Severe mental health issues including (but not limited to):
* Recent suicide attempt
* History of psychosis
* History of significant self-harm
* History of homicidal thoughts or actions
* History of violent behaviours sufficient to be considered a threat to others
* Acute eating disorder.
* Significant risk of absconding, or history of absconding
* Serious behavioural problems
* Significant use of drugs or alcohol
* History of sexual violence or sexual behaviour towards others
* Any significant interaction with the justice system or police
* Cognitive impairment that would interfere with treatment benefits
* Medical conditions that are not stable
* Severe medical conditions

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-07 (Estimated); Primary Completion 2014-07-30 (Actual); Study Completion 2014-07-30 (Actual)

PRIMARY OUTCOMES:
Post Traumatic Stress Disorder Symptom Severity | 4 Months
  PTSD symptom severity will be measured using the Child Post-Traumatic Stress Disorder Symptom Scale (CPSS)

SECONDARY OUTCOMES:
Quality of Life | 4 Months
  Quality of Life will be measured using the KidKindl, a 24 item self-report questionnaire.
Depression and Anxiety | 4 Months
  Depression and Anxiety will be measured using the Revised Children's Anxiety and Depression Scale (RCADS-Short Version)
Level of Attachment | 4 Months
  Level of Attachment will be measured using 5 secure attachment questions on a Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Farrel Greenspan, MC, Principal Investigator — University of Alberta
Locations (1):
- Be Brave Ranch, Ardrossan, Alberta, Canada